CLINICAL TRIAL: NCT06721884
Title: Herbal Evaluation Of Artemisia Annua For Small Intestinal Bacterial Overgrowth: A Phase I/II Triple-Masked, Placebo-Controlled Trial
Brief Title: Herbal Evaluation Of Artemisia Annua For Small Intestinal Bacterial Overgrowth
Acronym: HERBA-SIBO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: atelier temenos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RB71024
Record Dates: First submitted 2024-11-20; First posted 2024-12-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Small Intestinal Bacterial Overgrowth Syndrome (SIBO)
Keywords: randomized controlled trial; placebo; artemisia annua; SIBO; small intestinal bacterial overgrowth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artemisia annua (Experimental)
  Interventions: Dietary Supplement: Artemisia Annua Leaf
- Placebo (Placebo Comparator): We have chosen dried-leaf alfalfa of equal weight and dosing to the interventional product (5 grams, 15 caps, 5/am, 5/noon, 5/pm for the 4 weeks of the intervention period plus an additional 1 week dose escalation period to match the dosing of the Artemisia product). We have chosen this as a comparator in consultation with SIBO and herbal medicine content experts as alfalfa matches the texture and color of Artemisia annua and, in the doses used, will provide no meaningful amounts of FODMAPs or antimicrobial phytochemicals. The alfalfa will be sourced from Bulk Apotherapy, LCC, and encapsulated at the same facility as the Artemisia capsules. Containers of placebo capsules will be kept in a secured cabinet before being administered, under climate-controlled conditions, and checked weekly to ensure consistent ambient temperature.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Artemisia Annua Leaf — The intervention is Artecinua™ which is an organic Artemisia annua dried leaf powder in a vegan / kosher/ halal capsule. Artemisia annua L is classified as a 'generally regarded as safe' (GRAS) herb. Participants will be instructed to wean up to a full 5g dose by the following schedule.
  1. gram (3 caps) 1st day,
  2. grams (6 caps) 3/am, 3/pm, for the 3rd day,
  3. grams (9 caps) 3/am 3/noon 3/pm for the 5th day,
  4. grams (12 caps) 4/am, 4/noon, 4/pm for the 7th day,
  5. grams (15 caps) 5/am, 5/noon, 5/pm for rest of intervention period (4 weeks)
  Containers of ArtecinuaTM will be kept in a secured cabinet before being administered, under climate-controlled conditions, and checked weekly to ensure consistent ambient temperature.
  The justification of the 5g a day dosing is based on empiric experience and is in line with recommended dosages by the pharmacopeia of the People's Republic of China and has been previously used in clinical trials
  Arms: artemisia annua
Other: placebo — We have chosen dried-leaf alfalfa of equal weight and dosing to the interventional product (5 grams, 15 caps, 5/am, 5/noon, 5/pm for the 4 weeks of the intervention period plus an additional 1 week dose escalation period to match the dosing of the Artemisia product). We have chosen this as a comparator in consultation with SIBO and herbal medicine content experts as alfalfa matches the texture and color of Artemisia annua and, in the doses used, will provide no meaningful amounts of FODMAPs or antimicrobial phytochemicals. The alfalfa will be sourced from Bulk Apotherapy, LCC, and encapsulated at the same facility as the Artemisia capsules. Containers of placebo capsules will be kept in a secured cabinet before being administered, under climate-controlled conditions, and checked weekly to ensure consistent ambient temperature.
  Arms: Placebo

SUMMARY:
Small intestinal bacterial overgrowth (SIBO) can cause symptoms like bloating, stomach pain, and changes in bowel movements, significantly affecting quality of life. Many people with irritable bowel syndrome (IBS) also have SIBO, and there is growing recognition of how important it is to address this condition. Artemisia annua has shown potential in managing SIBO based on early reports and studies suggesting it can fight bacteria like *E. coli* and *Klebsiella*, which are linked to a type of SIBO that produces hydrogen gas.

This study aims to test if Artemisia annua is safe and well-tolerated for adults with hydrogen-type SIBO. Over five weeks, participants will take either 5 grams of dried Artemisia annua leaves or a placebo. Researchers will monitor safety through blood tests, vital signs, and adverse events, and they will assess symptom changes using questionnaires and breath tests.

The trial will include up to 32 participants from the Portland, Oregon area. Participants will be randomly assigned to treatment groups, and neither they, the researchers, nor the test administrators will know who is receiving the herb or the placebo. Results will be analyzed using standard statistical methods.

This study addresses the lack of research on herbal treatments for SIBO. If successful, the findings could lead to larger studies and help expand treatment options for people with SIBO.

DETAILED DESCRIPTION:
Background: Small intestinal bacterial overgrowth (SIBO) often leads to bloating, abdominal pain, and stool change, and has significant impacts on quality of life. There is a high prevalence of SIBO among irritable bowel syndrome patients in particular and a growing awareness in the medical community of the impact of this condition. Anecdotal reports indicate that Artemisia annua, traditionally used against malaria, has shown promise in individuals with SIBO and previous studies suggest it has antimicrobials effects against E. coli and Kelbsiella, the bacteria associated with the hydrogen subtype of SIBO. This protocol describes the design of a phase II triple blind placebo controlled trial aiming to evaluate the safety and tolerability of 5g a day of dried leaf Artemisia annua in treating adults with hydrogen subtype SIBO over a 5 week period. Secondary objectives include the impact on symptom severity and exploratory outcomes include hydrogen and methane gas response.

Methods: A triple-blind, placebo-controlled, parallel-arm trial will enroll up to 32 participants from the Portland Oregon metropolitan area. Participants will undergo two lactulose breath tests, biweekly blood tests, and regular symptom assessments. Randomization will be computer-generated, stratified by symptom severity, with adherence closely monitored. Outcomes will measure changes in laboratory toxicology indicators, vital statistics, adverse events, and symptom severity. Data will be analyzed using appropriate statistical tests with a significance level set at p<.05.

Discussion: This is a protocol for a phase II trial of Artemisia annua in individuals with hydrogen subtype SIBO. This study helps address the dearth of formal studies of herbal treatments for SIBO and the results could provide a basis for larger trials and contribute to broader treatment strategies for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* IBS-SSS score >175
* Meets North American Consensus criteria for H2 SIBO
* Willing to take Artecinua™ or placebo as a dietary supplement for 5 weeks
* Willing to have two lactulose breath tests and do the prep diet 24 hours before and fast overnight before the test
* Willing to have three blood drawstests and fast overnight before the draw
* Able to speak, read, and understand English
* Able to provide informed consent
* For individuals of child-bearing potential, willing to use an intrauterine device or two other concurrent forms of birth control to prevent pregnancy while enrolled

Exclusion Criteria:

* Use of antibiotic pharmaceuticals or supplements 14 days before baseline breath test
* Initiation of change in diet, medication, or supplement regime within 30 days
* Hospitalization within the past 3 months
* Women who are breastfeeding, pregnant, or planning pregnancy in the next 4 months
* Allergies to any of the ingredients in the study products.
* Individuals with chronic kidney or liver disease, cancer, colorectal disease and/or other rare disorders that at the discretion of the PI or Clinical *Investigator may impact their safety or confound trial results
* The use of any high-risk medications with narrow therapeutic indices metabolized by CYP450 enzymes: Warfarin (CYP2C9), Tacrolimus/Cyclosporine (CYP3A4), Efavirenz (CYP2B6), and Codeine (CYP2D6).
* Drugs requiring activation for efficacy: Clopidogrel (CYP2C19), Codeine (CYP2D6), and Tamoxifen (CYP2D6) (citations).
* GFR: <30 mL/min/1.73m²
* Hepatitis from any cause.
* Excessive alcohol use (> seven drinks/week in women and > fourteen in men).
* Hepatic (ALT, AST, bilirubin) and renal (creatinine, estimated GFR) parameters outside of normal range at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Complete blood count | 5 weeks
  RBC, WBC, platelets
Comprehensive metabolic profile | 5 weeks
  eGFR, electrolytes, BUN:Cr, AST, ALT, GGT, alkaline phosphatase, bilirubin
Vital sign measurement (heart rate) | 5 weeks
  bpm
Vital sign measurement (blood pressure) | 5 weeks
  mmHg
Vital sign measurement (temperature) | 5 weeks
  degrees F
Vital sign measurement (weight) | 5 weeks
  kg
Vital sign measurement (height) | 5 weeks
  meters
Vital sign measurement (body mass index) | 5 weeks
  weight (kg) / [height (m)]²
Adverse event monitoring | 5 weeks
  Adverse events
Quality of life | 5 weeks
  IBS-QoL

SECONDARY OUTCOMES:
Symptom severity | 5 weeks
  GI symptom severity (IBS-SSS)
Adequate relief | 5 weeks
  IBS-AR

OTHER OUTCOMES:
H2 gas response | 5 weeks
  H2 gas lactulose breath test. Day 0 to 35 difference measured by Δ baseline to 90 min in each test.
CH4 gas response | 5 weeks
  CH4 gas lactulose breath test. Day 0 to 35 difference measured by peak CH4 in each test.
Gas resolution | 5 weeks
  H2/CH4 lactulose breath test. Count of those with <20 ppm rise from baseline to 90 min H2 and <10 ppm absolute on CH4 by trial closeout.

CONTACTS AND LOCATIONS:
Locations (1):
- Helfgott Research Institute - National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No